CLINICAL TRIAL: NCT05070936
Title: Effect Of Vestibular Rehabilitation On Kinesiophobia, Quality Of Life, Dynamic Visual Acuity And Balance With Individuals Who Has Vestibular Hypofunction
Brief Title: The Effect Of Vestibular Rehabilitation On Kinesiophobia And Balance With Individuals Who Has Vestibular Hypofunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Ebru Sever, Specialist Physiotherapist, Istanbul Medipol University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-772.02-34270
Record Dates: First submitted 2021-10-06; First posted 2021-10-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Individuals With Vestibular Hypofunction; Individuals Between the Ages of 18-65
Keywords: Balance; Dynamic visual acuity; Kinesiophobia; Vestibular hypofunction; Vestibular rehabilitation
MeSH Terms: conditions — Kinesiophobia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- vestibular rehabilitation group (Other): Vestibular rehabilitation was performed. The following exercises were done with the patients: both sitting and standing gaze stabilization exercises, neck joint range of motion exercises, 20 minutes walks outside, walking backwards both open and closed eyes, and walking on tandem both open and closed eyes. Exercise program was applied for 8 weeks. Patients were observed in the hospital every two weeks. The exercises given in the session were given as home exercises, 3 times a day, for 10 repetitions.
  Interventions: Other: vestibular rehabilitation

INTERVENTIONS:
Other: vestibular rehabilitation — Vestibular rehabilitation consisted of a total of 4 sessions, rearranged every 15 days. These exercises were prepared gradually to increase the vestibulo-ocular reflex and vestibulospinal reflex. The following exercises were done with the patients: both sitting and standing gaze stabilization exercises, neck joint range of motion exercises, 20 minutes walks outside, walking backward both open-and-closed eyes, and walking in tandem with both open-and-closed eyes. The therapist gave the patients a home exercise program. It was emphasized that the exercises should be applied as 10 repetitions. After the session, the exercises shown to the patients were explained in written form and given as home exercises. They were also asked to do home exercises 3 times a day, 10 repetitions, for 15 days. Evaluation of the patients was done at the beginning of the first session and the 4th session. Thus, 3 separate exercise sessions and a home exercise program were applied to the patients.

SUMMARY:
Vestibular hypofunction is a disease which emerge through a partial or total loss on a vestibular organ or vestibular nerve. It can be seen unilateral or bilateral. Aim of the study is to examine effects of vestibular rehabilitation on kinesiophobia, quality of life, dynamic vision acuity and balance. The study was conducted with patients diagnosed with vestibular hypofunction. 30 patients who are in the ages between 18 and 65 have participated in the study. Exercise programs has given to patients to do at home. Patients were observed every two weeks in the hospital. The following exercises were done with the patients: both sitting and standing gaze stabilization exercises, neck joint range of motion exercises, 20 minutes walks outside, walking backwards both open and closed eyes, and walking on tandem both open and closed eyes. Exercise program was applied for 8 weeks. Before and after the treatment, Tampa Kinesiophobia Scale, World Health Organization Quality of Life Scale-Short form in Turkish, Dynamic Visual Acuity Test, Balance Tests, Unterberger Test, Visual Analog Scale to measure dizziness and fatigue, for verticality and horizontality perception Subjective Visual Vertical and Subjective Visual Horizontal tests have been applied. As a result of the study, statistical correlations have been found except semi-tandem posture test with eyes open and Romberg's test both with eyes open and closed. It can be said that vestibular rehabilitation has improved quality of life, balance, dynamic vision acuity and overcame kinesiophobia on the patients.

DETAILED DESCRIPTION:
Vestibular rehabilitation consisted of a total of 4 sessions, rearranged every 15 days. These exercises were prepared gradually to increase the vestibulo-ocular reflex and vestibulospinal reflex. The following exercises were done with the patients: both sitting and standing gaze stabilization exercises, neck joint range of motion exercises, 20 minutes walks outside, walking backward both open-and-closed eyes, and walking in tandem with both open-and-closed eyes. The therapist gave the patients a home exercise program. It was emphasized that the exercises should be applied as 10 repetitions. After the session, the exercises shown to the patients were explained in written form and given as home exercises. They were also asked to do home exercises 3 times a day, 10 repetitions, for 15 days. Evaluation of the patients was done at the beginning of the first session and the 4th session. Thus, 3 separate exercise sessions and a home exercise program were applied to the patients.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with vestibular hypofunction diagnosed by videonystagmography test
* Patients aged between 18-65 years.

Exclusion Criteria:

* Patients with visual impairment and neurological involvement
* Individuals with wavy vertigo
* Ataxia, or other lesions causing oscillopsia
* Dementia
* Patients with severely limited mobility and unable to walk without using a walker, cane, or orthosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2021-04-02 (Actual)

PRIMARY OUTCOMES:
Before and After Tampa Kinesiophobia Scale Values | 8 Weeks
  It was determined that there was a statistically significant difference between the before and after measurement values of the Tampa kinesiophobia scale dimensions.

SECONDARY OUTCOMES:
World Health Organization Quality of Life Scale-Short form Before and After Values | 8 Weeks
  It was determined that there was a statistically significant difference between the pre- and post-measurement values of the World Health Organization Quality of Life Scale-Short form dimensions.
: Results of Tandem Stance Test, Subjective Visual Vertical and Subjective Visual Horizontal Tests, Dizziness Severity and Dynamic Visual Acuity Parameters | 8 Weeks
  Improvements were observed in the tandem stance test eyes open/eyes closed test Subjective Visual Vertical and Subjective Visual Horizontal test scores on sitting, hard and soft surfaces were found to be statistically significant. The mean vertigo severity (VAS) decreased from 7.15±1.36 to 1.06±2.02.It was found that there was a statistically significant difference between the pre- and post-measurement values of the visual acuity test score.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Sever, master, Principal Investigator — master student; Z.Candan Algun, professor, Study Director — head of physical medicine and rehabilitation department
Locations (1):
- Güneşli Erdem Hastanesi, Bağcılar, Güneşli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No